CLINICAL TRIAL: NCT01398995
Title: To Consider the Effect of the Timing of a Reduction in Basal Insulin Infusion Rate to 50% of Normal Prior to Exercise on Glycaemic Control in People With Type 1 Diabetes Treated With CSII
Brief Title: Managing Insulin Pumps for Exercise (Study 2)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was terminated due to elevated levels of hypoglycaemia
Sponsor: Buckinghamshire Healthcare NHS Trust (Other)
Collaborators: Animas Corporation (Industry)
Responsible Party: Denise Watson, Research and Development Manager, Buckinghamshire Hospitals NHS Trust
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: RXQ404
Record Dates: First submitted 2011-07-20; First posted 2011-07-21 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Exercise; continuous subcutaneous insulin infusion
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 90 minutes (Experimental): Basal insulin infusion reduced to 50% of normal 90 minutes prior to exercise
  Interventions: Other: Reduction of basal insulin infusion to 50% of normal
- 60 minutes (Experimental): Basal insulin infusion reduced to 50% of normal 60 minutes prior to exercise
  Interventions: Other: Reduction of basal insulin infusion to 50% of normal
- 30 minutes (Experimental): Basal insulin infusion reduced to normal 30 minutes prior to exercise
  Interventions: Other: Reduction of basal insulin infusion to 50% of normal
- Start (Experimental): Basal insulin infusion reduced to 50% of normal at the start of exercise
  Interventions: Other: Reduction of basal insulin infusion to 50% of normal

INTERVENTIONS:
Other: Reduction of basal insulin infusion to 50% of normal — Each participant in this cross-over trial will participate in the 4 arms of the trial. They will be presented with the four conditions in randomised order - reducing their basal insulin infusion rate to 50% of normal at the four time points specified. A comparison will be made between the conditions.

SUMMARY:
People with Type 1 Diabetes Mellitus (T1DM) like to take part in sport and exercise, but problems with metabolism and blood glucose control can make this difficult. Some people with T1DM administer their insulin via an insulin pump, also know as continuous subcutaneous insulin infusion (CSII) therapy, in which a background or basal level of insulin is constantly infused under the skin by a special pump, with bolus doses of insulin given to accompany food. Clinical experience suggests that this may be particularly useful for managing diabetes for exercise, but there is limited experimental evidence to support this. The aim of this research , which is divided into three parts, is to investigate the hypothesis that the physiological response to sub-maximal (moderate) exercise of a person with type 1 diabetes treated with CSII, can be made to approximate more closely to the physiological response of a healthy individual by a prior reduction of their basal insulin infusion rate. Evidence from children demonstrates that reducing the basal insulin infusion rate to 50% of normal at the beginning of exercise can reduce rates of low blood glucose (hypoglycaemia) during exercise. However, reducing the insulin infusion rate will not have an immediate effect on levels of insulin in the body, and evidence from adults suggests that the level of insulin in the bloodstream at the start of exercise is an important factor in whether hypoglycaemia develops during exercise. This suggests that reducing the basal insulin infusion rate some time before exercise may be useful. The aim of this study is to compare the effect of a basal insulin reduction on blood glucose levels between visits when this reduction is made at the start of exercise, 30 minutes before, 60 minutes before and 90 minutes before. The null hypothesis to be tested is that there is no difference between these conditions.

DETAILED DESCRIPTION:
Participants recruited will have type 1 diabetes treated with CSII. Each participant will be required to attend on 5 separate occasions. The first visit can take place at any time of day. At this first visit formal, written consent will be obtained for participation in the trial. Following this an assessment will be made of VO2 MAX(maximal oxygen uptake during exercise) using the Balke-Ware treadmill protocol. Once this is finished the first visit will be completed.

The other 4 visits will all take place 2 hours following a lunch containing 60 grams of carbohydrate. Advice will be given about how this can be achieved. On arrival a cannula will be inserted in the dorsum of a hand and blood samples taken. The hand will be armed to allow the taking of arterialised blood samples. Further blood samples will be taken after 30, 60 and 90 minutes and then exercise will commence. Participants will be asked to reduce their basal insulin infusion rate to 50% of usual either immediately after the cannula has been inserted or 30 minutes later (1 hour prior to exercise), 60 minutes later (30 minutes prior to exercise) or 90 minutes later (at the start of exercise). These four conditions will be presented to each participant in a randomised order. Participants will exercise for 60 minutes at 50% VO2 MAX on an electronically braked cycle ergometer. At the end of exercise a set of blood samples will be taken. Participants will then rest for 30 minutes and a final set of blood samples will be taken. After this the cannula will be removed and the study visit will be complete. A snack will be offered.

In the event of hypoglycaemia identified on point of care testing a blood sample will be taken for laboratory confirmation. Participants will be given 15 grams of carbohydrate but permitted to continue exercising unless they feel that the exercise has become significantly more difficult, they feel unwell or the investigator has any concerns. Participants will be given 15 grams of rapid acting carbohydrate, repeated every 10-15 minutes until blood glucose levels rise above 4mmol/l.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged between 18 and 65 years
* Diagnosed with Type 1 diabetes mellitus
* Treated with CSII for at least 3 months
* Exercises regularly for more than 1 hour per week

Exclusion Criteria:

* People with any one of the following complications of diabetes:

  * stage 2+ diabetic retinopathy
  * renal impairment (with creatinine >150micromol/l)
  * known history or symptoms of cardiovascular disease
  * foot ulceration
  * peripheral vascular disease
* Known pregnancy or breastfeeding
* Untreated or unstable respiratory disease
* Known hypoglycaemia unawareness
* Treatment with drugs known to interfere with glucose metabolism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Comparison of glucose excursion (change in blood glucose) between baseline and the end of exercise between the four conditions. | Samples taken on arrival and at the end of exercise

SECONDARY OUTCOMES:
Comparison between the four conditions of change in blood glucose levels between baseline and the beginning of exercise, and between the beginning and end of exercise. | Samples taken at baseline, beginning and end of exercise
Levels of NEFA and lactate will be compared between the four conditions | Samples will be taken at the 6 time points detailed below
  Samples will be taken in each condition at baseline (90 minutes prior to exercise), after 30 minutes (60 minutes prior to exercise), after 60 minutes (30 minutes prior to exercise), after 90 minutes (at the start of exercise), after 150 minutes (at the end of 1 hour of exercise) and at 180 minutes (30 minutes after the end of exercise)
Correlation between levels of NEFA and lactate and blood glucose will be considered. | Samples will be taken at the time points detailed below
  Samples will be taken in each condition at baseline (90 minutes prior to exercise), after 30 minutes (60 minutes prior to exercise), after 60 minutes (30 minutes prior to exercise), after 90 minutes (at the start of exercise), after 150 minutes (at the end of 1 hour of exercise) and at 180 minutes (30 minutes after the end of exercise)
Ratio of respiratory quotient (RQ) at the beginning of exercise to RQ at the end of exercise compared between the four conditions. | Breath by breath data will be recorded for 2 minutes at the start and the end of the exercise period

CONTACTS AND LOCATIONS:
Overall Officials: Ian W Gallen, MD FRCP, Principal Investigator — Buckinghamshire Healthcare NHS Trust
Locations (1):
- Wycombe Hospital, High Wycombe, Buckinghamshire, United Kingdom